CLINICAL TRIAL: NCT00941356
Title: A Single Center, Double-Blind, Randomized, Placebo-Controlled Study Evaluating the Efficacy of Bio-K+ Cl-1285® In the Nasal Decolonization of Methicillin Resistant Staphylococcus Aureus (MRSA) Carrier Patients
Brief Title: Evaluation of the Efficacy of Bio-K+ Cl-1285® In the Nasal Decolonization of Methicillin Resistant Staphylococcus Aureus (MRSA) Carrier Patients
Acronym: MRSA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to recruit patients to continue on with the study.
Sponsor: Bio-K Plus International Inc. (Industry)
Collaborators: Centre Hospitalier Pierre-Le Gardeur (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL1285-MRSA-M03
Record Dates: First submitted 2009-01-15; First posted 2009-07-17 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: MRSA Colonization
Keywords: MRSA nasal colonisation; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Bio-K+ CL1285 contains 50 billion of live bacteria
  Interventions: Dietary Supplement: Bio-K+ CL1285
- 2 (Placebo Comparator): placebo devoid of bacteria
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bio-K+ CL1285 — 2 capsules per day before breakfast
  Other Names: Bio-K+ CL1285(R) Extra Strength
  Arms: 1
Dietary Supplement: Placebo — 2 capsules per day before breakfast
  Arms: 2

SUMMARY:
Trial Objectives:

Primary objective:

* To evaluate the efficacy of Bio-K+CL1285® in patients with Methicillin-Resistant S. aureus (MRSA) nasal colonization by comparing the MRSA decolonization following either Bio-K+CL1285® or placebo treatment.

Secondary objective:

* To evaluate the safety profile of Bio-K+CL1285®.

DETAILED DESCRIPTION:
Study Design:

Double-blind, randomized (1:1 randomization), placebo-controlled, single center Canadian study.

Patients will be randomly assigned to one of the two study products. A randomization schedule will be generated by the sponsor for each participating centre. This schedule will link patient identification numbers to one of the two study products allocated at random. The schedule will be prepared on a 1:1 randomization ratio.

The study products will be labelled with the patient identification number. Patients have to be randomized in the order in which they qualify from the screening phase for inclusion in the study.

Patients withdrawn from the study retain their patient number if already given. New patients must always be allotted a new identification number (PIN).

Study Duration:

The duration of patient participation in the study will be between 22 and 23 days. The overall duration of the study is expected to be approximately 10 months; with subject recruitment proposed to start in March 2009, the last follow-up visit is expected in May 2010. The actual overall study duration or subject recruitment period may vary.

Number of Sites (inside and outside of Canada):

One center in the province of Quebec will be involved in the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients having ≥18 years of age
* Women of child bearing capacity who are not pregnant at the moment of screening (Pregnancy test done on-site) and agree to use an acceptable form of birth control for the duration of the study (e.g. condom, oral contraceptives, etc.) are allowed to participate.
* Patients must have nasal MRSA colonization confirmed with MRSA positive culture as assessed during the screening visit without any clinical signs or symptoms of infection.
* Laboratory test results within the normal ranges.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients treated for nasal MRSA decolonization in the last 6 months;
* Current infection with MRSA;
* Ongoing or active infection;
* Daily probiotic/ fermented milk or Yogurt use;
* Known to have shown a previous reaction, including anaphylaxis, to any substance in composition of the study agent (capsules);
* Ongoing or recent use of antibiotics in the 30 days prior to the study agent administration;
* Pregnancy, breastfeeding;
* Regular use of nasal agents;
* Uncontrolled intercurrent illness, including situations that would limit compliance with study requirements;
* Patients with open wounds
* Immunosuppressive therapy or any health condition causing inmunosuppression (Including Haematological malignancies, AIDS);
* Ostomized patients, parenteral nutrition users;
* Patients with current vascular access (catheter) or planned to have installed a vascular access (catheter) or any prosthesis during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Frequency of subjects with MRSA decolonization | 21 days

SECONDARY OUTCOMES:
To evaluate the secondary effects (incidence rate of non-serious ans serious adverse events)associated to the administration of the study product | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr Pierre-Jean PM Maziade, MD, Principal Investigator — Pierre Le Gardeur Hospital
Locations (1):
- Pierre Le Gardeur Hospital, Terrebonne, Quebec, Canada